CLINICAL TRIAL: NCT05610540
Title: Patient Preference and Visual Quality With Contralateral Synergy Versus Panoptix
Status: Completed | Type: Observational
Sponsor: Bucci Laser Vision Institute (Other)
Responsible Party: Sponsor
Other Study IDs: FAB-1274
Record Dates: First submitted 2022-10-31; First posted 2022-11-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: IOL; Cataract; Patient Satisfaction
MeSH Terms: conditions — Cataract; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: TECNIS Synergy IOL — Implanted in one eye
Device: AcrySof PanOptix Trifocal IOL — Implanted in one eye

SUMMARY:
The goal of this study is to compare the visual quality and patient preference of the Synergy IOL versus the PanOptix IOL when one of each lens is placed in the same patient.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation have been planned for both eyes
* Desire to mitigate postoperative presbyopia with implantation of Synergy IOL in one eye and PanOptix Trifocal IOL in the opposite eye

Exclusion Criteria:

* Any vision-limiting problems (e.g., corneal, retinal, infection) which can potentially limit post-operative visual performance
* Any ocular condition or trauma that is not resolved, stable, or would compromise the well-being of the subject

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females, aged 40 and older, with bilateral cataracts
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction - subjective questionnaire | 3 months to 18 months after cataract surgery
  Subjective questionnaire explores the frequency and need for glasses for various visual functions at distance, intermediate, and near and overall satisfaction of visual function without glasses
Visual Acuity at Distance | 3 months to 18 months after cataract surgery
  Uncorrected and best corrected visual acuities measured at distance
Visual Acuity at Intermediate | 3 months to 18 months after cataract surgery
  Uncorrected and best corrected visual acuities measured at intermediate
Visual Acuity at Near | 3 months to 18 months after cataract surgery
  Uncorrected and best corrected visual acuities measured at near

CONTACTS AND LOCATIONS:
Locations (1):
- Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania, United States